CLINICAL TRIAL: NCT03831503
Title: A Phase 1 Study of INO-A002 in Healthy Dengue Virus-naive Adults
Brief Title: A Study of INO-A002 in Healthy Dengue Virus-naive Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 832135
Record Dates: First submitted 2019-01-29; First posted 2019-02-05 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: This study will adhere to a dose escalation scheme. There are five cohorts for Study ZIKA-dMAb 01. Participants (n=6 per cohort) will be administered INO-A002 at four dose levels: 0.5, 1, 2, and 4 mg DNA/dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (5):
- Cohort A - 0.5mg (Experimental): Participants (n=6 per cohort) will be administered 1 injection (Day 0) of INO-A002 at 0.5 mg DNA/dose. Inoculation will be administered as 0.5 ml IM injection followed by electroporation with the CELLECTRA® 2000 device.
  Interventions: Biological: INO-A002; Device: CELLECTRA® 2000; Device: Dengue Fever Antibodies (IgG)
- Cohort B - 1mg (Experimental): Participants (n=6 per cohort) will be administered 1 injection (Day 0) of INO-A002 at 1 mg DNA/dose. Inoculation will be administered as 1 ml IM injection followed by electroporation with the CELLECTRA® 2000 device.
  Interventions: Biological: INO-A002; Device: CELLECTRA® 2000; Device: Dengue Fever Antibodies (IgG)
- Cohort C - 2mg (Experimental): Participants (n=6 per cohort) will be administered 2 injections (Day 0 and Day 3) of INO-A002 at 2 mg DNA/dose. Inoculation will be administered as 1 ml IM injection followed by electroporation with the CELLECTRA® 2000 device.
  Interventions: Biological: INO-A002; Device: CELLECTRA® 2000; Device: Dengue Fever Antibodies (IgG)
- Cohort D - 4mg (Experimental): Participants (n=6 per cohort) will be administered 2 injections (Day 0 and Day 3) of INO-A002 at 4 mg DNA/dose. Inoculation will be administered as 1 ml IM injection followed by electroporation with the CELLECTRA® 2000 device.
  Interventions: Biological: INO-A002; Device: CELLECTRA® 2000; Device: Dengue Fever Antibodies (IgG)
- Cohort E - 4mg Side Port (Experimental): Participants (n=6 per cohort) will be administered 2 injections (Day 0 and Day 3) of INO-A002 at 4 mg DNA/dose. Inoculation will be administered as 1 ml IM injection followed by electroporation with the CELLECTRA® 2000 device with Side Port needle.
  Interventions: Biological: INO-A002; Device: CELLECTRA® 2000; Device: Dengue Fever Antibodies (IgG)

INTERVENTIONS:
Biological: INO-A002 — Participants will receive one or two 1 ml IM injections (in different arms) into the deltoid region at day 0 (all groups), and in addition on day 3 (in the 2 mg and 4 mg cohorts).
Device: CELLECTRA® 2000 — Inoculation will be followed by electroporation with the CELLECTRA® 2000 device.
Device: Dengue Fever Antibodies (IgG) — To determine if the subject is Dengue seronegative at baseline

SUMMARY:
Phase 1, open label, single center, dose escalation study to evaluate the safety, tolerability and pharmacokinetic profile of dMAb-ZK190 following delivery of INO-A002 with Hylenex® recombinant delivered IM followed by EP in healthy adult Dengue naïve volunteers ages 18-60 years.

DETAILED DESCRIPTION:
This is a Phase 1, open label, single center, dose escalation study to evaluate the safety, tolerability and pharmacokinetic profile of dMAb-ZK190 following delivery of INO-A002 with Hylenex® recombinant delivered IM followed by EP in healthy adult Dengue naïve volunteers ages 18-60 years.

The study will apply a 3+3 design such that 3 additional subjects will be enrolled into the cohort if one DLT (Section 7.3.1) is observed in one out of the first 3 subjects dosed during the 28-day period of safety and PK assessment. If no additional DLT is observed in 3 additional subjects (i.e., 1 DLT in 6 total subjects), dosing will proceed to the subsequent cohort. However, if any additional DLT occurs (i.e., >1 DLT in 6 total subjects), then that dose will be deemed not tolerated and the prior dose will be considered the maximum tolerated dose (MTD).

ELIGIBILITY:
1. Age 18-60 years;
2. Able to provide consent to participate and having signed an Informed Consent Form (ICF);
3. Able and willing to comply with all study procedures;
4. Body mass index (BMI) between 20 and 30, inclusive
5. Screening laboratory must be within normal limits or have only Grade 0-1 findings;
6. Normal screening ECG or screening ECG with no clinically significant findings;
7. Women of child-bearing potential agree to use medically effective contraception (oral contraception, barrier methods, spermicide with barrier methods, etc.) or have a partner who is sterile from enrollment to 6 months following the last injection, or have a partner who is medically unable to induce pregnancy.
8. Sexually active men who are considered sexually fertile must agree to use either a barrier method of contraception during the study, and agree to continue the use for at least 6 months following the last injection, or have a partner who is permanently sterile or is medically unable to become pregnant;
9. No history of clinically significant immunosuppressive or autoimmune disease. Individuals with HIV infection who have been virologically suppressed for more than 1 year and with current CD4 cell count entry greater than 500 cells/ul will be allowed into the study.
10. No history of dengue virus vaccination or illness; no history of yellow fever vaccination.
11. Dengue seronegative at baseline by screening laboratory evaluation
12. Not currently or within the previous 4 weeks taking immunosuppressive agents (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or prednisone at a dose less than 10 mg/day or steroid dose-equivalent).

Exclusion Criteria:

1. Administration of an investigational compound either currently or within 30 days of first dose;
2. Previous receipt of an investigational product for the treatment or prevention of Zika virus except if participant is verified to have received placebo;
3. Administration of any vaccine within 4 weeks of first dose;
4. Administration of any monoclonal or polyclonal antibody product within 4 weeks of the first dose
5. Administration of any blood product within 3 months of first dose;
6. Pregnancy or breast feeding or plans to become pregnant during the course of the study;
7. Positive serologic result for dengue virus (any serotype) or history of receipt of either dengue virus or yellow fever virus vaccination at any time in the past;
8. Positive serologic test for hepatitis B surface antigen (HBsAg); or any potentially communicable infectious disease as determined by the Principal Investigator or Medical Monitor;
9. Positive serologic test for hepatitis C (exception: successful treatment with confirmation of sustained virologic response);
10. Baseline evidence of kidney disease as measured by creatinine greater than 1.5 (CKD Stage II or greater);
11. Baseline screening lab(s) with Grade 2 or higher abnormality, except for Grade 2 creatinine;
12. Chronic liver disease or cirrhosis;
13. Immunosuppressive illness including hematologic malignancy, history of solid organ or bone marrow transplantation;
14. Current or anticipated concomitant immunosuppressive therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or prednisone at a dose greater than 10 mg/day or steroid dose-equivalent);
15. Current or anticipated treatment with TNF-α inhibitors such as infliximab, adalimumab, etanercept;
16. Prior major surgery or any radiation therapy within 4 weeks of group assignment;
17. Any pre-excitation syndromes, e.g., Wolff-Parkinson-White syndrome;
18. Presence of a cardiac pacemaker or automatic implantable cardioverter defibrillator (AICD)
19. Fewer than two acceptable sites available for IM injection and EP considering the deltoid and anterolateral quadriceps muscles. The following are unacceptable sites:

    * Tattoos, keloids or hypertrophic scars located within 2 cm of intended administration site;
    * Implantable-Cardioverter-defibrillator (ICD) or pacemaker (to prevent a life-threatening arrhythmia) that is located ipsilateral to the deltoid injection site (unless deemed acceptable by a cardiologist);
    * Any metal implants or implantable medical device within the electroporation site.
20. Prisoner or participants who are compulsorily detained (involuntary incarceration) for treatment of either a physical or psychiatric illness;
21. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements or assessment of immunologic endpoints; or
22. Not willing to allow storage and future use of samples for Zika virus related research
23. Any illness or condition that in the opinion of the investigator may affect the safety of the participant or the evaluation of any study endpoint.
24. Participants who plan to travel within 6 months of INO-A002 administration to a geographic location where DENV or ZIKV are currently active.
25. Participants with known bleeding diatheses or that are using blood thinners for 30 days before study enrollment including warfarin, heparin, Clopidogrel, Apixaban (Eliquis), Dabigatran (Pradaxa), Edoxaban (Savaysa), Rivaroxaban (Xarelto). The use of low dose aspirin (81 mg daily) will be acceptable.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of escalating doses of INO-A002 with Hylenex® administered IM followed by electroporation with the CELLECTRA® 2000 device in healthy adult volunteers. | 52 weeks
  Safety will be assessed by monitoring the frequency and severity of adverse events utilizing the "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" with labs assessed as per site normal values.
Evaluate the tolerability of escalating doses of INO-A002 with Hylenex® administered IM followed by electroporation with the CELLECTRA® 2000 device in healthy adult volunteers. | 10 minutes
  Pain will be assessed by administration (i.e., injection) site reactions (frequency and severity) and visual analogue scale (VAS) scores.
Determine the maximum serum concentration (Cmax) of the monoclonal antibody dMAb-ZK190 in the serum upon administration of INO-A002 with Hylenex® delivered IM followed by electroporation. | 52 weeks
  The maximum serum concentration (Cmax) assessment will be performed by the analysis of dMAb-ZK190 levels at baseline; days 1, 3, 7 and at weeks 2, 3, 4, 5, 6, 8, 12, 16, 24 and 52. Serum concentration in micrograms/mL will be used as the measurement scale.
Determine the minimum serum concentration (Cmin) of the monoclonal antibody dMAb-ZK190 in the serum upon administration of INO-A002 with Hylenex® delivered IM followed by electroporation. | 52 weeks
  The minimum serum concentration (Cmin) assessment will be performed by the analysis of dMAb-ZK190 levels at baseline; days 1, 3, 7 and at weeks 2, 3, 4, 5, 6, 8, 12, 16, 24 and 52. Serum concentration in micrograms/mL will be used as the measurement scale.
Determine the Area Under the Curve (AUC0-t) of the monoclonal antibody dMAb-ZK190 in the serum upon administration of INO-A002 with Hylenex® delivered IM followed by electroporation | 52 weeks
  The Area Under the Curve (AUC0-t) will be performed by the analysis of dMAb-ZK190 levels at baseline; days 1, 3, 7 and at weeks 2, 3, 4, 5, 6, 8, 12, 16, 24 and 52. The Area Under the Curve (AUC0-t) against time will be calculated using the trapezoidal method.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Tebas, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States